CLINICAL TRIAL: NCT03020940
Title: 100000 Cases Real World Research of the Safety and Efficacy Revaluation of Cefuroxime Axetil Dispersible Tablets After Listing
Brief Title: The Clinical Trial of Cefuroxime Axetil Dispersible Tablets
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: FM-P5-2016072201-1
Record Dates: First submitted 2017-01-06; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-08

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases | interventions — cefuroxime axetil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cefuroxime Axetil Dispersible Tablets — Oral. This product can be taken orally, can also be added to the amount of warm water after mixing evenly.
  Adult general 0.25g (one time), 2 times a day, the general course of treatment for 5 to 10 days.
  Severe Infection or suspected pneumonia, a 0.5g (once 2), 2 times a day; general urinary tract infection, a Times a 0.125g (one and a half tablets), 2 times a day; for patients with no complications of gonorrhea recommended dose of 1g (4 Tablets), a single taking.
  Children generally a dose of 0.125g (one-half tablets), 2 times a day; for less than two years of age in the middle ear Inflammatory patients, a 0.125g (one half tablets), 2 times a day; for greater than two years of otitis media patients, one Times a 0.25g (one time), 2 times a day; more than 12 years of age in children, the same dose for adults

SUMMARY:
1. National, large-scale, standardized, standardized, real-world research;
2. Prospective, single - arm open, non - interventional, registration, multi - center clinical study;
3. in the use of cefuroxime axetil dispersible tablets in the hospital, according to the principle of voluntary selection of 200;
4. registration of the use of cefuroxime axetil dispersion tablets patients;
5. Target sample size of 100,000 cases;
6. Exemption from informed consent for ethical review applications;
7. Antibiotic drug safety re-evaluation of large data.

DETAILED DESCRIPTION:
Research purposes

1. To evaluate the safety of cefuroxime axetil dispersible tablets in the real world of the widely used population,

   Rare or even very rare, new, unanticipated adverse reactions, while revealing adverse reactions

   Should be susceptible to risk factors and susceptible populations.
2. To evaluate the efficacy of cefuroxime axetil dispersible tablets in the treatment of the relevant site of infection, including

   Including empirical therapy and targeted therapy, to further evaluate the widespread use of cefuroxime dispersible tablets

   The validity of the crowd in the real world.
3. To investigate the clinical application of cefuroxime axetil dispersible tablets for the safety management of drug use.

   Clinical management should provide more clinical clues and basis.
4. For the relevant treatment areas of guidance and consensus revision, clinical pathway design provides a reference.
5. To further improve the safety of cefuroxime axetil dispersion tablets level, the basic medical security capabilities and Market vitality.

Study end point

1. The main study endpoint:

   * Security;
   * Effectiveness.
2. Secondary study endpoint:

   * Extensive use of population characteristics;
   * Clinical drug characteristics;
   * Appropriate characteristics of the crowd;
   * Adverse reactions susceptible population characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Prescription of cefuroxime axetil dispersible tablets in patients

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prescription of cefuroxime axetil dispersible tablets in patients
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Bacterial clearance | 1 to 14 days after the use of Cefuroxime Axetil Dispersible Tablets，
  1.clear 2.Assume purge 3.Not cleared 4.Assume not cleared 5.Partially cleared 6.replace 7.Re-infection 8.Colonization 9.Can not be evaluated

IPD SHARING:
Plan to Share IPD: Undecided